CLINICAL TRIAL: NCT03481790
Title: The Effect of Orally Administered Iron-saturated Lactoferrin on Systemic Iron Homeostasis in Pregnant Women Suffering From Iron Deficiency and Iron Deficiency Anaemia
Brief Title: Lactoferrin Versus Ferrous Sulphate for Treatment of Iron Deficiency Anaemia During Pregnancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Khaled Mohamed Balsha, principal investigator, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AinShams Maternity Hospital
Record Dates: First submitted 2018-03-12; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Iron Deficiency Anemia of Pregnancy
Keywords: iron deficiency anemia of pregnancy - lactoferrin
MeSH Terms: interventions — Lactoferrin; ferrous sulfate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactoferrin (Experimental): 100mg of bovine lactoferrin (Pravotin sachets, Hygint, Egypt) twice a day.
  Interventions: Drug: Lactoferrin
- ferrous sulphate + folic acid (vitamin B9) (Experimental): 150mg of dried ferrous sulphate + folic acid (vitamin B9) 0.50mg (Ferrofol, E.I.P.I.C.O, Egypt) three capsules per day.
  Interventions: Drug: ferrous sulphate + folic acid (vitamin B9)

INTERVENTIONS:
Drug: Lactoferrin — (Pravotin sachets, Hygint, Egypt): 100 mg in 1/4 glass of water before meals twice a day for 4 weeks.
  Other Names: Pravotin; MamyVital
  Arms: Lactoferrin
Drug: ferrous sulphate + folic acid (vitamin B9) — (Ferrofol capsules, Eipico, Egypt): Dried ferrous sulphate 150 mg + Folic acid (Vitamin B9) 150 mg at least 1 hour before or 2 hours after meals three times a day for 4 weeks.
  Other Names: Ferrofol
  Arms: ferrous sulphate + folic acid (vitamin B9)

SUMMARY:
This study evaluates the efficacy and tolerability of lactoferrin in contrast to ferrous sulphate in the context of iron deficiency anemia with pregnancy.

Half of participants will receive lactoferrin, while the other half will receive ferrous sulphate.

DETAILED DESCRIPTION:
Lactoferrin and Ferrous sulfate are used to treat iron deficiency anemia in pregnancy.

Ferrous sulphate is the most commonly used treatment for iron deficiency anemia.

Lactoferrin is a new generation oral iron that has long been recognized as a member of the transferrin family of proteins and an important regulator of the levels of free iron in the body fluids and has the ability to enhance iron binding. Preliminary evidence suggests that lactoferrin may represent a promising new strategy for oral iron replacement.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with single fetus
* Hb count < 11g/dL
* ferritin level < 12 ng/dL
* Gestational age (14 - 30 weeks)

Exclusion Criteria:

* Associated chronic medical disorder (CKD, liver disease, peptic ulcer and chronic blood loss).
* Associated bleeding disorder
* Anaemia requiring blood tranfusion (Hb < 7g/dL)
* Hypersensitivity to iron preparations
* Haemoglobinopathies (G6PD, thalassemias, sickle cell disease)

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Hemoglobin (Hb) level. | 4 weeks
  to be measured before and after treatment.

SECONDARY OUTCOMES:
serum ferritin level. | 4 weeks
  to be measured before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mamdouh, Study Director — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No